CLINICAL TRIAL: NCT01363245
Title: Effectiveness of Smoking-cessation Interventions for Urban Hospital Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHART NYU; 1U01HL10522901 (Other Grant/Funding Number: NHLBI); 3U01HL105229-03S2 (NIH)
Record Dates: First submitted 2011-01-31; First posted 2011-06-01 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Smoking Cessation
Keywords: cost effectiveness; behavioral health counseling
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hospital phone counseling (Experimental): multisession telephone counseling by hospital/study's smoking cessation staff
  Interventions: Behavioral: Telephone Counseling
- Fax-to-quit (Active Comparator): Faxed referral to the state Quitline, which will then perform phone outreach as per Quitline protocol
  Interventions: Behavioral: Fax-to-quit

INTERVENTIONS:
Behavioral: Telephone Counseling — Telephone counseling: 7 calls over 6 weeks
  Arms: Hospital phone counseling
Behavioral: Fax-to-quit — referral to state smoking cessation 'quitline' for counseling - 1 call over 2 weeks
  Arms: Fax-to-quit

SUMMARY:
The investigators plan to compare the effectiveness and cost effectiveness of an inpatient smoking cessation intervention for all smokers hospitalized at two urban public hospitals.

DETAILED DESCRIPTION:
Our sites are: Bellevue Hospital Center (a New York City public hospital) and the Manhattan campus of the VA New York Harbor Healthcare System. During hospitalization, all smokers will receive usual care. At the time of discharge, patients will be randomized to one of two arms: multisession telephone counseling by their hospital's smoking cessation staff, or faxed referral to the state Quitline (which will then perform phone outreach as per Quitline protocol). All patients enrolled in the study will receive nicotine replacement therapy.

The primary aims are:

Aim 1: To compare the effectiveness of the intervention (proactive multisession telephone counseling by in-hospital staff) versus control ('fax-to-quit' Quitline referral).

Aim 2: To evaluate and compare the cost-effectiveness of these interventions from a societal perspective and from a payer perspective.

The secondary aims are:

Secondary Aim 1: To compare outcomes by race/ethnicity, immigrant status, inpatient diagnosis, and location of patient hospitalization Secondary Aim 2: To compare outcomes of the interventions at 6 and 12 months post-discharge Secondary Aim 3: To compare biochemically-verified abstinence rates at 6 months post-discharge Secondary Aim 4: To compare cessation outcomes between those who are known HIV-seropositive and those who are not, and explore possible mediators of cessation in HIV-seropositive patients

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* smoked tobacco during the prior 30 days
* have an active phone number
* provide consent in English, Spanish or Mandarin

Exclusion Criteria:

* Patients will be excluded if they use only smokeless tobacco or products such as betel (since there is not yet efficacy data for treating use of these tobacco products in the inpatient setting)
* are pregnant or breastfeeding
* are discharged to an institution (e.g. jail/prison, nursing home, long-term psychiatric facility).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1618 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness of counseling intervention vs. control intervention on smoking cessation rates of participants enrolled in study | 4 yrs
  To compare the effectiveness of a phone counseling intervention (proactive multisession telephone counseling by in-hospital staff) versus control intervention ('fax-to-quit' Quitline referral)

SECONDARY OUTCOMES:
Comparison of cessation outcomes by sociodemographic subgroups | 4yrs
  To compare smoking abstinence rates by race/ethnicity, immigrant status, inpatient diagnosis, and location of patient hospitalization
Comparison of cessation rates at 6 and 12 months post-discharge | 4yrs
  To compare smoking abstinence rates in the two arms at 6 months and 12 months post-discharge
Comparison of biochemically-verified smoking cessation | 4 years
  To compare rates of biochemically-verified smoking abstinence measured at 6 months post-discharge
Comparison of cessation outcomes between participants who are HIV-seropositive vs. those who are not | 2 years
  To compare cessation outcomes between those who are known HIV-seropositive and those who are not, and explore possible mediators of cessation in HIV-seropositive patients.
Cost Effectiveness comparison of two smoking cessation interventions. | 4 yrs
  Evaluate and compare the cost-effectiveness of these interventions from a societal perspective and from a payor perspective. Our hypotheses are that the intervention will have incremental cost-effectiveness ratios consistent with current standards of healthcare value in the United States.

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Sherman, MD, MPH, Principal Investigator — NYU School of Medicine
Locations (2):
- United States (2):
  - VA New York Harbor Healthcare System, New York, New York
  - Bellevue Hospital Center, New York, New York

REFERENCES:
- [Derived] Triant VA, Grossman E, Rigotti NA, Ramachandran R, Regan S, Sherman SE, Richter KP, Tindle HA, Harrington KF. Impact of Smoking Cessation Interventions Initiated During Hospitalization Among HIV-Infected Smokers. Nicotine Tob Res. 2020 Jun 12;22(7):1170-1177. doi: 10.1093/ntr/ntz168. PMID 31687769
- [Derived] Cody GR, Wang B, Link AR, Sherman SE. Characteristics of Urban Inpatient Smokers With and Without Chronic Pain: Foundations for Targeted Cessation Programs. Subst Use Misuse. 2019;54(7):1138-1145. doi: 10.1080/10826084.2018.1563186. Epub 2019 Feb 1. PMID 30706753
- [Derived] Sherman SE, Link AR, Rogers ES, Krebs P, Ladapo JA, Shelley DR, Fang Y, Wang B, Grossman E. Smoking-Cessation Interventions for Urban Hospital Patients: A Randomized Comparative Effectiveness Trial. Am J Prev Med. 2016 Oct;51(4):566-77. doi: 10.1016/j.amepre.2016.06.023. PMID 27647057
- [Derived] Duffy SA, Cummins SE, Fellows JL, Harrington KF, Kirby C, Rogers E, Scheuermann TS, Tindle HA, Waltje AH; Consortium of Hospitals Advancing Research on Tobacco (CHART). Fidelity monitoring across the seven studies in the Consortium of Hospitals Advancing Research on Tobacco (CHART). Tob Induc Dis. 2015 Sep 3;13(1):29. doi: 10.1186/s12971-015-0056-5. eCollection 2015. PMID 26336372
- [Derived] Grossman E, Shelley D, Braithwaite RS, Lobach I, Goffin A, Rogers E, Sherman S. Effectiveness of smoking-cessation interventions for urban hospital patients: study protocol for a randomized controlled trial. Trials. 2012 Aug 1;13:126. doi: 10.1186/1745-6215-13-126. PMID 22852878